CLINICAL TRIAL: NCT05450471
Title: Effectiveness of Endonasal Polymeric Implant in the Treatment of Chronic Eosinophilic and Central Compartment Rhinosinusitis: a Randomized Controlled Trial
Brief Title: Effectiveness of Endonasal Polymeric Implant for Chronic Rhinosinusitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luiz Eduardo Florio Junior, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USPStudy
Record Dates: First submitted 2022-01-14; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Rhinosinusitis Chronic
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-lactide and trimethynele carbonate Terpolymers polymer implant (Experimental): The polymer implant will be placed in the ethmoidal region, at the same time that the nasal endoscopic examination will be performed. The polymer in this study is biocompatible. The polymers will be made in the biomaterials laboratory located at the Pontifical Catholic University of São Paulo (PUC-SP), located in the city of Sorocaba-SP. Polymers will be provided free of charge for the study.
  Interventions: Drug: Corticosteroid Topical
- Placebo polymer implant (Placebo Comparator): Placebo polymer implant
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Corticosteroid Topical — The L-lactide and trimethynele carbonate (TCM) Terpolymers polymer implant will be placed in the ethmoidal region, at the same time that the nasal endoscopic examination will be performed.
  Arms: L-lactide and trimethynele carbonate Terpolymers polymer implant
Other: Placebo — Placebo
  Arms: Placebo polymer implant

SUMMARY:
Objective: The objective of this study is to evaluate a steroid-embedded Terpolymers polymer implant of L-lactide and trimethynele carbonate (TCM) at the level of disease control in patients with eosinophilic and central compartment chronic rhinosinusitis (CRS) after placement of the endonasal device, compared to a control group (placebo). The secondary objectives of this study are to assess comfort, perception of improvement and satisfaction, as well as adverse events.

Methods: A randomized controlled trial will be carried out, with a blinded participant, therapist and evaluator. Patients over 18 years of age, with chronic rhinosinusitis (CRS) who have already undergone endoscopic sinus surgery (CENS), but who do not have the disease under control and, therefore, with an indication for a new CENS, will be selected. Participants will come from the otorhinolaryngology outpatient clinic of the academic and public service of the University of São Paulo - USP. Eligible patients will receive either the Terpolymers L-lactide and trimethynele carbonate (TCM) polymer implant placement or the placebo polymer. The primary outcome will be the control of the symptoms of chronic uncontrolled rhinosinusitis that will be evaluated through the NOSE Questionnaire, a nasal endoscopic evaluation based on the Lund-Kennedy criteria and the SNOT-22 Questionnaire. The sample size calculation was performed based on a difference between the intervention and placebo groups of 30% for cases that achieved disease control, resulting in a sample of 36 participants (18 in each group). Data will be analyzed using mixed linear models.

ELIGIBILITY:
Inclusion Criteria:

- Patients with chronic rhinosinusitis undergoing endoscopic sinus surgery, but who do not have the disease under control. The uncontrolled disease and its respective classification regarding the degree of the disease will be carried out through 3 assessments: 1) Nose Obstruction Symptom Evaluation Questionnaire (NOSE) validated version in Portuguese; 2) nasal endoscopic evaluation; and, 3) Sino Nasal Outcome Test Questionnaire (SNOT-22). Through the NOSE questionnaire, the patient's disease will be classified as "Controlled", "Partially Controlled" or "Uncontrolled (Uncontrolled)". Any variation in the endoscopic evaluation score based on the Lund-Kennedy Criteria will be considered an alteration. And for the SNOT-22 Questionnaire, changes will be considered when the total score varies by at least 11 points. Patients who present these 3 alterations will be considered to have the 'uncontrolled disease' and, therefore, will be eligible for the study.

Exclusion Criteria:

* Patients with malformations, trauma and/or tumors in the nasal and paranasal sinuses will be excluded;
* Patients with a history of recent nasal surgery up to 6 months previously, with glaucoma and cataracts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Nasal Obstruction | Day 15 after intervention
  Nasal Obstruction, Sistemic medication and Endoscopy (NOSE) questionnaire. NOSE is a method of evaluating the clinical control of chronic rhinosinusitis and is based on the evaluation of three aspects: nasal obstruction, nasal endoscopy and the need for systemic medication (antibiotics or steroids).
  The NOSE questionnaire consists of five questions concerning subjective assessment of the nasal obstruction within the past month. Each question can be answered usinga 5-point Likert scale from"0"(not a problem) up to"4"(severe problems with breathing). After addition of allitem values and multiplying the raw score with 5, severity of the patient's complaints can be scaled to range from 0 to 100. A score of 0 indicates no obstructivenasal problems and a score of 100 implies severe problems.
Nasal Endoscopic Evaluation | Day 15 after intervention
  The nasal endoscopic evaluation will be performed under topical anesthesia, with a rigid endoscope (4mm, 0° and/or 45°; Karl Storz) and its classification will be based on the Lund - Kennedy criteria. For this evaluation, each nostril is examined separately and three possible characteristics may be present, they are: polyps, nasal mucosa edema and/or secretion. For each evaluated characteristic, a score from 0 to 2 is assigned. For the evaluation of polyps, the score is applied as follows: 0=absent; 1=restricted to the middle meatus; and, 2=extension to nasal cavity. For the evaluation of nasal mucosa edema, the score is applied as follows: 0=absent; 1=mild or moderate edema; and 2= polypoid degeneration. For the evaluation of secretion, the score is applied as follows: 0=absent; 1=hyaline secretion; and, 2=mucopurulent or thick secretion.
Sino Nasal Outcome Test | Day 15 after intervention
  Sino Nasal Outcome Test (SNOT-22) The SNOT-22 Questionnaire is a modification of the SNOT-20, with 2 additional items on nasal obstruction and problems with smell and taste. The questionnaire assesses 22 items related to nasal symptoms that can impact the patient's personal and social life. Each item can get a score ranging from 0 (least possible problem) to 5 (greatest possible problem). Thus, this questionnaire has a final score that can range from 0 to 110 points. In this study, a significant clinical improvement will be considered when there is at least a variation of 11 points from one assessment to another.23 The validity and reliability of the SNOT-22 have already been previously tested in Portuguese.

SECONDARY OUTCOMES:
Morning serum level of cortisol, albumin and serum globulin | Day 15 after intervention
  blood test
Morning serum level of cortisol, albumin and serum globulin | Day 60 after intervention
  blood test
ACTH - adrenocorticotropic hormone | Day 15 and 60 aftern intervention
  blood test
ACTH - adrenocorticotropic hormone | Day 15 after intervention
  blood test
Complete blood count | Day 60 after intervention
  A complete blood count (CBC) is a blood test used to evaluate your overall health and detect a wide range of disorders, including anemia, infection and leukemia.
  A complete blood count test measures several components and features of your blood, including:
  Red blood cells, which carry oxygen White blood cells, which fight infection Hemoglobin, the oxygen-carrying protein in red blood cells Hematocrit, the proportion of red blood cells to the fluid component, or plasma, in your blood Platelets, which help with blood clotting
total and serum IgE (blood test) | Day 15 after intervention
  blood test
total and serum IgE (blood test) | Day 60 after intervention
  blood test
Cortisol level in 24-hour urine | Day 15 after intervention
  urine test
Cortisol level in 24-hour urine | Day 60 after intervention
  urine test
Intraocular pressure profile - IOP | Day 15 after intervention
  ophthalmologic assessment - fluid overload test and the lens by slit lamp examination
Intraocular pressure profile - IOP | Day 60 after intervention
  ophthalmologic assessment - fluid overload test and the lens by slit lamp examination
Patient comfort | Day 15 after intervention
  self-reported on an analog scale from 0 to 100, where 0 indicates very uncomfortable and 100 indicates very comfortable
Patient comfort | Day 60 after intervention
  self-reported on an analog scale from 0 to 100, where 0 indicates very uncomfortable and 100 indicates very comfortable
Patient self-reported perception of improvement and satisfaction with the implant | Day 15 after intervention
  Measured on an analog scale from 0 to 100, where 0 indicates no change in symptoms and dissatisfaction, and 100 indicates resolved symptoms and satisfaction
Patient self-reported perception of improvement and satisfaction with the implant | Day 60 after intervention
  Measured on an analog scale from 0 to 100, where 0 indicates no change in symptoms and dissatisfaction, and 100 indicates resolved symptoms and satisfaction
Adverse events | Day 15 after intervention
  Adverse events will be measured through changes in blood and urine tests and also on a self-reported basis.
Adverse events | Day 60 after intervention
  Adverse events will be measured through changes in blood and urine tests and also on a self-reported basis.
Nasal Obstruction | Day 45 after intervention
  Nasal Obstruction, Sistemic medication and Endoscopy (NOSE) questionnaire. NOSE is a method of evaluating the clinical control of chronic rhinosinusitis and is based on the evaluation of three aspects: nasal obstruction, nasal endoscopy and the need for systemic medication (antibiotics or steroids).
  The NOSE questionnaire consists of five questions concerning subjective assessment of the nasal obstruction within the past month. Each question can be answered usinga 5-point Likert scale from"0"(not a problem) up to"4"(severe problems with breathing). After addition of allitem values and multiplying the raw score with 5, severity of the patient's complaints can be scaled to range from 0 to 100. A score of 0 indicates no obstructivenasal problems and a score of 100 implies severe problems.
Nasal Obstruction | Day 90 after intervention
  Nasal Obstruction, Sistemic medication and Endoscopy (NOSE) questionnaire. NOSE is a method of evaluating the clinical control of chronic rhinosinusitis and is based on the evaluation of three aspects: nasal obstruction, nasal endoscopy and the need for systemic medication (antibiotics or steroids).
  The NOSE questionnaire consists of five questions concerning subjective assessment of the nasal obstruction within the past month. Each question can be answered usinga 5-point Likert scale from"0"(not a problem) up to"4"(severe problems with breathing). After addition of allitem values and multiplying the raw score with 5, severity of the patient's complaints can be scaled to range from 0 to 100. A score of 0 indicates no obstructivenasal problems and a score of 100 implies severe problems.
Nasal Endoscopic Evaluation | Day 45 after intervention
  The nasal endoscopic evaluation will be performed under topical anesthesia, with a rigid endoscope (4mm, 0° and/or 45°; Karl Storz) and its classification will be based on the Lund - Kennedy criteria. For this evaluation, each nostril is examined separately and three possible characteristics may be present, they are: polyps, nasal mucosa edema and/or secretion. For each evaluated characteristic, a score from 0 to 2 is assigned. For the evaluation of polyps, the score is applied as follows: 0=absent; 1=restricted to the middle meatus; and, 2=extension to nasal cavity. For the evaluation of nasal mucosa edema, the score is applied as follows: 0=absent; 1=mild or moderate edema; and 2= polypoid degeneration. For the evaluation of secretion, the score is applied as follows: 0=absent; 1=hyaline secretion; and, 2=mucopurulent or thick secretion.
Nasal Endoscopic Evaluation | Day 90 after intervention
  The nasal endoscopic evaluation will be performed under topical anesthesia, with a rigid endoscope (4mm, 0° and/or 45°; Karl Storz) and its classification will be based on the Lund - Kennedy criteria. For this evaluation, each nostril is examined separately and three possible characteristics may be present, they are: polyps, nasal mucosa edema and/or secretion. For each evaluated characteristic, a score from 0 to 2 is assigned. For the evaluation of polyps, the score is applied as follows: 0=absent; 1=restricted to the middle meatus; and, 2=extension to nasal cavity. For the evaluation of nasal mucosa edema, the score is applied as follows: 0=absent; 1=mild or moderate edema; and 2= polypoid degeneration. For the evaluation of secretion, the score is applied as follows: 0=absent; 1=hyaline secretion; and, 2=mucopurulent or thick secretion.
Sino Nasal Outcome Test | Day 45 after intervention
  Sino Nasal Outcome Test (SNOT-22) The SNOT-22 Questionnaire is a modification of the SNOT-20, with 2 additional items on nasal obstruction and problems with smell and taste. The questionnaire assesses 22 items related to nasal symptoms that can impact the patient's personal and social life. Each item can get a score ranging from 0 (least possible problem) to 5 (greatest possible problem). Thus, this questionnaire has a final score that can range from 0 to 110 points. In this study, a significant clinical improvement will be considered when there is at least a variation of 11 points from one assessment to another.23 The validity and reliability of the SNOT-22 have already been previously tested in Portuguese.
Sino Nasal Outcome Test | Day 90 after intervention
  Sino Nasal Outcome Test (SNOT-22) The SNOT-22 Questionnaire is a modification of the SNOT-20, with 2 additional items on nasal obstruction and problems with smell and taste. The questionnaire assesses 22 items related to nasal symptoms that can impact the patient's personal and social life. Each item can get a score ranging from 0 (least possible problem) to 5 (greatest possible problem). Thus, this questionnaire has a final score that can range from 0 to 110 points. In this study, a significant clinical improvement will be considered when there is at least a variation of 11 points from one assessment to another.23 The validity and reliability of the SNOT-22 have already been previously tested in Portuguese.

CONTACTS AND LOCATIONS:
Locations (1):
- Luiz Eduardo Flório Junior, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided